CLINICAL TRIAL: NCT03337113
Title: Working Memory Training Combined With Transcranial Magnetic Stimulation in Smokers: 2x2 Factorial Study
Brief Title: Working Memory Training Combined With Transcranial Magnetic Stimulation in Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: Brown University (Other); Butler Hospital (Other)
Responsible Party: Principal Investigator, William Lechner. PhD, Assistant Professor, Kent State University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1705-003
Record Dates: First submitted 2017-10-25; First posted 2017-11-08 (Actual); Results first posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Transcranial Magnetic Stimulation; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: A 2x2 factorial model will include four groups (Working Memory Training [WMT] + repetitive Transcranial Magnetic Stimulation ]rTMS], sham WMT+rTMS, WMT+sham TMS, and sham WMT+sham rTMS) capable of isolating independent and combined effects of WMT and rTMS on the primary outcome variables.
Who Masked: Participant, Care Provider
Masking Description: The participant will be prevented from having knowledge of the interventions assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- WMT + rTMS (Experimental): WMT + rTMS is the Working Memory Training + repetitive Transcranial Magnetic Stimulation arm. Both conditions are active.
  Interventions: Other: Working Memory Training; Device: repetitive Transcranial Magnetic Stimulation
- Sham WMT + rTMS (Active Comparator): Sham WMT + rTMS is the sham Working Memory Training + repetitive Transcranial Magnetic Stimulation arm. This condition isolates the effects of rTMS. WMT is inactive.
  Interventions: Other: Sham Working Memory Training; Device: repetitive Transcranial Magnetic Stimulation
- WMT + sham rTMS (Active Comparator): WMT + sham rTMS is the Working Memory Training + sham repetitive Transcranial Magnetic Stimulation arm. This condition isolates the effects of WMT. rTMS is inactive.
  Interventions: Other: Working Memory Training; Device: Sham repetitive Transcranial Magnetic Stimulation
- Sham WMT + sham rTMS (Sham Comparator): sham WMT + sham rTMS is the sham Working Memory Training + sham repetitive Transcranial Magnetic Stimulation arm. Both are inactive in this arm.
  Interventions: Other: Sham Working Memory Training; Device: Sham repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Other: Working Memory Training — The Working Memory Training condition: This condition will include 30 sessions across 4 weeks (10 remote sessions prior to initiation of the rTMS stimulation, and 20 lab sessions on rTMS stimulation days). Participants will complete three distinct WM tasks in each session: a visuospatial WM task, a backward digit span task, and a letter span task. In the training condition, the difficulty level of all three WM tasks will be automatically adjusted on a trial-by-trial basis. An identical protocol and software have demonstrated efficacy in increasing WM capacity, and this improvement in WM predicts reduction in addictive behavior.
  Other Names: Executive Function Training
  Arms: WMT + rTMS; WMT + sham rTMS
Other: Sham Working Memory Training — In the Sham WMT condition, the difficulty level of the WM tasks will not be adjusted; instead it will remain at the initial easy level throughout each task (i.e., three items in each sequence). All other aspects of the condition are identical to the active WMT condition.
  Other Names: Sham Executive Function Training
  Arms: Sham WMT + rTMS; Sham WMT + sham rTMS
Device: repetitive Transcranial Magnetic Stimulation — The rTMS Condition: rTMS will be delivered with a Magstim Rapid2 system using Magstim Air Film Coils. rTMS pulses will be delivered at 10 Hz (100% resting motor threshold, RMT) in 40, 5 second trains, with 15 second inter-train interval, for a total of 2000 pulses per session. Active or sham rTMS will be applied over the left DLPFC; corresponding with the standard "F3" location on scalp (F3=left frontal lobe, location #3 for electrode placement using international 10-20 system for scalp measurements). Five consecutive daily sessions will occur on two consecutive weeks, for a total of 10 sessions. RMT, defined as the amount of energy required to induce movement in the contralateral abducer pollicis brevis in at least 50% of stimulations, will be assessed on first day of application.
  Other Names: Neuromodulation
  Arms: Sham WMT + rTMS; WMT + rTMS
Device: Sham repetitive Transcranial Magnetic Stimulation — Sham rTMS will be identical to active treatment, with the exception that mu-metal plates attached to the sham coil block the magnetic field while providing a sensation of stimulation.
  Other Names: Sham Neuromodulation
  Arms: Sham WMT + sham rTMS; WMT + sham rTMS

SUMMARY:
Smoking remains the leading cause of preventable death in the United States, and current first-line treatments leave the majority of tobacco dependent individuals unable to quit. The inability to quit despite motivation to do so, is thought to result in part, from self-control failure. Working memory (WM) deficits contribute to imbalanced self-control and allow automatic impulses to drive behavior. Thus, WM plays a critical role in addictive behavior, and is particularly relevant to smoking. Indeed, a strong link between WM and smoking has been established in the literature; most notably, degree of WM impairment and deficits in activation in associated brain regions predict time to relapse, and WM moderates the relationship between craving and relapse. Given these insights, researchers have been examining interventions that may target WM including WM training (WMT) and repetitive Transcranial Magnetic Stimulation (rTMS). WMT involves taxing this executive function repeatedly over time and has shown positive preliminary results in improving measures of self-control and reducing consumption of addictive substances. Similarly, rTMS, a non-invasive brain stimulation procedure that stimulates neuronal tissues and increases cortical excitability, has been shown to increase WM capacity and reduce craving and consumption of several addictive substances including nicotine. While these interventions have demonstrated initial promise in affecting addictive behaviors, the magnitude and durability of their effects may be limited. Recently, researchers have posited - but not yet empirically tested - that WMT administered in combination with rTMS may result in an additive or supra-additive effect in treating addictive processes. This is highly significant; the clinical utility of rTMS over current first line treatments may be limited if factors with potential to enhance its effectiveness are not examined. Given these recent advances in the literature, the primary objective of the proposed study is to evaluate the individual and combined effects of Working Memory (WM) training and repetitive Transcranial Magnetic Stimulation (rTMS) on WM performance and smoking behaviors as well as critical mediators of these effects. These aims will be examined in a sample of tobacco dependent adults (N=130) utilizing a 2x2 factorial experimental design including four groups (WMT+rTMS, sham WMT+rTMS, WMT+sham TMS, and sham WMT+sham rTMS) capable of isolating independent and combined effects of WMT and rTMS.

DETAILED DESCRIPTION:
SPECIFIC AIMS Smoking remains the leading cause of preventable death in the U.S. Current first line treatments leave approximately 70% of tobacco dependent individuals unsuccessful in their attempt to quit. Specifically, only 5-30% of those who initiate treatment, including intensive first-line interventions, are able to maintain abstinence for one or more years. The inability to quit despite motivation to do so is thought to result, in part, from self-control failure and can be understood within the framework of dual process models of addiction. Dual process models view vulnerability to tobacco dependence as the relative balance between automatic impulses and control processes orchestrated through the interplay of multiple executive function. Working memory (WM) is an executive function associated with updating information to solve immediate problems, and achieve current goals. WM is a key cognitive process underlying the regulatory control component of dual process models and is involved in the initiation, maintenance, and relapse stages of tobacco dependence. Most notably, deficits in WM performance and activation in associated brain regions predict time to relapse and strong WM has been shown to reduce the effect of craving on the ability to resist smoking. Given this relationship, individuals with tobacco dependence are likely to benefit from interventions that strengthen WM. Recently, several studies have demonstrated that increasing WM capacity through WM training (WMT) is associated with positive outcomes in several populations with substance use or impulse control disorders. Specifically, studies have demonstrated that WMT is associated with decreased: delay discounting in substance users, weight re-gain after a weight loss program, and alcohol use in heavy drinkers.

A second emerging innovation in the treatment of addictions is repetitive Transcranial Magnetic Stimulation (rTMS), a procedure which sends magnetic pulses through the scalp to stimulate neuronal tissue resulting in observed changes in neuronal plasticity and striatal dopamine. rTMS has now demonstrated positive effects in several substance use disorders including nicotine, alcohol, and stimulant dependence. This procedure has been shown to be effective in reducing smoking urges in abstinent as well as satiated smokers and to reduce cigarette consumption. While promising results for this treatment have been demonstrated, the size and durability of the therapeutic effect may be limited. Additionally, the mechanism by which rTMS exerts positive effects on smoking outcomes is unknown. Recently it has been posited that changes in WM performance resulting from rTMS may be the key pathway to its observed effects on smoking related outcomes, and furthermore that WMT administered in close temporal precedence to rTMS may result in an additive or supra-additive effect in treating addictive processes. However, these hypotheses have not been tested to date despite their importance for understanding and improving the clinical impact of these emerging therapeutic modalities for treating addictive behaviors. Interventions with the ability to effectively target self-control processes fill in a critical gap in currently available treatment options.

The primary objective of the proposed study is to evaluate the potential for improved effects and examine mediating pathways of WMT in combination with rTMS on a laboratory based smoking task and neuropsychological measures of WM performance. These aims will be examined in a sample of tobacco dependent adults (N=130) utilizing a 2x2 factorial design including four groups (WMT+rTMS, sham WMT+rTMS, WMT+sham TMS, and sham WMT+sham rTMS) capable of isolating independent and combined effects of WMT and rTMS. The study will include a baseline laboratory assessment, 10 WMT sessions over two weeks, followed by 10 days of WMT immediately preceding and following brain stimulation sessions (10 Hz rTMS, 2000 pulses per session, applied to left DLPFC). Neurocognitive and psychological mediators will be assessed between baseline and final laboratory assessment. Lastly, a follow-up assessment will occur one-month after the final laboratory visit. The proposed study will test the following Specific Aims:

Aim 1: To test the potential for improved effects of combining WMT with rTMS on smoking behaviors as compared to the independent effects of either condition alone. Hypothesis: Single active conditions (WMT+sham rTMS and sham WMT+rTMS) will result in significant increases in time to lapse on an analogue task as compared to the double sham condition (sham WMT+sham rTMS), and the WMT+rTMS condition will result in significant increases in time to lapse as compared to the single active conditions.

Aim 2: To test the potential for improved effects of combining WMT with rTMS on WM performance.

Hypothesis: WMT + rTMS will result in significant increases in WM performance as compared to all other conditions, including the additive increases in conditions outlined in Aim 1.

Aim 3: To test mediating pathways of the effects rTMS on smoking behaviors including changes in craving, mood, and WM performance. Hypothesis: The direct effect of rTMS on smoking outcomes will be mediated by gains in WM performance, and this effect will be largest in the WMT+rTMS condition.

ELIGIBILITY:
Inclusion Criteria:

* meet safety guidelines for application of rTMS
* be 18-60 years of age
* have smoked cigarettes regularly for at least one year
* currently smoke at least 10 cigarettes per day
* have a carbon monoxide (CO) level >10 ppm
* currently use no other nicotine products regularly

Exclusion Criteria:

* meet criteria for current alcohol or substance dependence
* have a current affective disorder (depression, dysthymia, or mania) or psychotic symptoms
* are currently pregnant or lactating, or intend to become pregnant
* have a health condition for which rTMS is contraindicated

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William V Lechner, Ph.D., Principal Investigator — Kent State University
Locations (2):
- United States (2):
  - Brown University, Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared.

REFERENCES:
- [Derived] Lechner WV, Philip NS, Kahler CW, Houben K, Tirrell E, Carpenter LL. Combined Working Memory Training and Transcranial Magnetic Stimulation Demonstrates Low Feasibility and Potentially Worse Outcomes on Delay to Smoking and Cognitive Tasks: A Randomized 2 x 2 Factorial Design Pilot and Feasibility Study. Nicotine Tob Res. 2022 Nov 12;24(12):1871-1880. doi: 10.1093/ntr/ntac183. PMID 35907262

RESULTS

PARTICIPANT FLOW:
Groups:
- WMT + rTMS: WMT + rTMS is the Working Memory Training + repetitive Transcranial Magnetic Stimulation arm. Both conditions are active.
  Working Memory Training: The Working Memory Training condition: This condition will include 30 sessions across 4 weeks (10 remote sessions prior to initiation of the rTMS stimulation, and 20 lab sessions on rTMS stimulation days). Participants will complete three distinct WM tasks in each session: a visuospatial WM task, a backward digit span task, and a letter span task. In the training condition, the difficulty level of all three WM tasks will be automatically adjusted on a trial-by-trial basis.
  repetitive Transcranial Magnetic Stimulation: The rTMS Condition: rTMS will be delivered with a Magstim Rapid2 system using Magstim Air Film Coils. rTMS pulses will be delivered at 10 Hz (100% resting motor threshold, RMT) in 40, 5 second trains, with 15 second inter-train interval, for a total of 2000 pulses per session. Active or sham rTMS will be applied over the left DLPFC; corresponding with the standard "F3" location on scalp (F3=left frontal lobe, location #3 for electrode placement using international 10-20 system for scalp measurements). Five consecutive daily sessions will occur on two consecutive weeks, for a total of 10 sessions. RMT, defined as the amount of energy required to induce movement in the contralateral abducer pollicis brevis in at least 50% of stimulations, will be assessed on first day of application.
Period: Overall Study
Arm/Group | WMT + rTMS | Sham WMT + rTMS | WMT + Sham rTMS | Sham WMT + Sham rTMS
Started | 13 | 12 | 12 | 13
Completed | 12 | 9 | 11 | 11
Not Completed | 1 | 3 | 1 | 2
Not completed — Adverse Event | 1 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WMT + rTMS | Sham WMT + rTMS | WMT + Sham rTMS | Sham WMT + Sham rTMS | Total
Number analyzed (Participants) | 12 | 9 | 11 | 11 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (10.45) | 44.77 (8.05) | 45.72 (9.23) | 40.36 (9.88) | 43.25 (9.43)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 4 | 3 | 3 | 4 | 14
  Gender: Male | 7 | 6 | 8 | 7 | 28
  Gender: Does not Identify as Male or Female | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race / Ethnicity: Non-Hispanic White | 11 | 9 | 9 | 8 | 37
  Race / Ethnicity: Non-Hispanic Black | 0 | 0 | 1 | 1 | 2
  Race / Ethnicity: Non-Hispanic Multiracial | 1 | 0 | 1 | 1 | 3
  Race / Ethnicity: Hispanic White | 0 | 0 | 0 | 1 | 1
Education (12 years or less) [Count of Participants; unit: Participants]
  12 years or less | 3 | 3 | 4 | 1 | 11
  more than 12 years | 9 | 6 | 7 | 10 | 32
Employment [Count of Participants; unit: Participants]
  Not working | 7 | 3 | 2 | 5 | 17
  working at least part time | 5 | 6 | 9 | 6 | 26
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 17.16 (7.48) | 18.33 (7.93) | 22.27 (8.02) | 17.54 (5.41) | 18.81 (7.30)
Fagerstrom Test for Cigarette Dependence (FTCD) [Mean (Standard Deviation); unit: units on a scale] — Total score range = 0 - 10.
  Higher scores indicate higher cigarette dependence.
  units on a scale | 6.58 (1.88) | 6.56 (1.66) | 6.27 (1.00) | 6.00 (2.00) | 6.35 (1.64)
General Cigarette Craving (past 24 hrs) [Mean (Standard Deviation); unit: units on a scale] — Cigarette Craving in the 24 hours preceding baseline assessment.
  Score range = 0 - 3.
  Higher score indicates higher craving.
  units on a scale | 1.83 (1.03) | 1.67 (1.00) | 1.82 (.75) | 1.45 (.82) | 1.70 (.88)
Age started smoking (years) [Mean (Standard Deviation); unit: years] | 14.25 (2.09) | 14.11 (3.14) | 12.63 (4.31) | 14.36 (2.41) | 13.83 (3.06)

OUTCOME MEASURES:

1. Primary Outcome: Time to Lapse on a Smoking Lapse Analogue Task
Description: The Delay to Smoking Analogue Task is a behavioral choice paradigm that is sensitive to smoking medication effects in which participants earn monetary rewards for delaying initiation of cigarette smoking in 5-minute increments over a 50-minute period, following 3-hours of observed smoking deprivation. Range = 0 - 50 minutes. Higher scores indicate better ability to delay smoking.
Time Frame: an average of 30 days after baseline
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | WMT + rTMS | Sham WMT + rTMS | WMT + Sham rTMS | Sham WMT + Sham rTMS
Number analyzed (Participants) | 9 | 7 | 11 | 8
minutes | 16.11 (24.21) | 38.0 (18.65) | 26.36 (25.40) | 15.25 (18.49)

2. Primary Outcome: Working Memory Performance 1
Description: NIH Examiner N-back score. The minimum value is 0 and maximum is 90, higher scores indicate a better outcome. Calculated change scores are presented (outcome score at day 30 minus baseline score).
Time Frame: Change from baseline score to score at 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WMT + rTMS | Sham WMT + rTMS | WMT + Sham rTMS | Sham WMT + Sham rTMS
Number analyzed (Participants) | 12 | 9 | 11 | 10
units on a scale | 7.08 (6.58) | 4.11 (7.08) | 3.73 (4.96) | 4.67 (7.01)

3. Primary Outcome: Working Memory Performance 2
Description: NIH Examiner Dot Counting Task score. The minimum total score is 0 and the maximum score is 27, higher scores indicate a better outcome. Calculated change scores are presented (outcome score at day 30 minus baseline score).
Time Frame: Change from baseline score to score at 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WMT + rTMS | Sham WMT + rTMS | WMT + Sham rTMS | Sham WMT + Sham rTMS
Number analyzed (Participants) | 12 | 9 | 11 | 10
units on a scale | 1.75 (1.96) | 1.44 (7.16) | 0.73 (5.48) | 0.80 (3.94)

4. Primary Outcome: Working Memory Performance 3
Description: Mean End Level Score on Maastricht University Working Memory Tasks. For each scale (i.e. visuospatial, back-digit, and letter-sequencing) the minimum total is 3 and the maximum is 15, higher scores indicate a better outcome.
Time Frame: Change from baseline score to score at 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WMT + rTMS | Sham WMT + rTMS | WMT + Sham rTMS | Sham WMT + Sham rTMS
Number analyzed (Participants) | 12 | 8 | 11 | 11
units on a scale
  Maastricht Visuospatial | 1.33 (.776) | 1.00 (1.60) | 1.00 (1.18) | .636 (1.29)
  Maastricht Back digit | 1.00 (2.52) | 1.62 (1.41) | 3.73 (2.69) | .910 (2.70)
  Maastricht Letter-Sequencing | 3.25 (2.26) | 2.38 (3.38) | 2.0 (3.0) | 1.82 (2.32)

5. Primary Outcome: Cigarette Consumption
Description: Self reported number of cigarettes smoked daily
Time Frame: throughout 60 day study participation, cigarettes per day assessed at outcome reported
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | WMT + rTMS | Sham WMT + rTMS | WMT + Sham rTMS | Sham WMT + Sham rTMS
Number analyzed (Participants) | 12 | 9 | 11 | 11
cigarettes per day | 16.00 (10.82) | 15.33 (9.0) | 17.36 (9.89) | 15.72 (11.28)

6. Secondary Outcome: Delay Discounting
Description: Discounting Rate on the Monetary Choice Questionnaire, assessed by k (log transformed). Individuals made hypothetical choices between smaller immediate rewards (e.g. $11 today) and larger delayed rewards (e.g. $30 in 7 days) at varying levels of hyperbolic-like discounting. Overall temporal discounting function (k) was assessed; larger values indicate steeper discounting which reflects a worse outcome.
  Total score range = 0 - 0.25.
Time Frame: Change from baseline score to score at 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WMT + rTMS | Sham WMT + rTMS | WMT + Sham rTMS | Sham WMT + Sham rTMS
Number analyzed (Participants) | 12 | 9 | 11 | 11
units on a scale | .131 (.377) | .202 (.316) | -.178 (3.06) | -.053 (.552)

7. Secondary Outcome: Cigarette Demand
Description: Demand characteristics on the Cigarette Purchase Task. Demand sensitivity indicates sensitivity to change in price, with higher values reflecting higher sensitivity to the monetary reinforcer rather than the substance, thus higher scores reflect a better outcome. Score range = 0 - .100.
Time Frame: Change from baseline score to score at 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | WMT + rTMS | Sham WMT + rTMS | WMT + Sham rTMS | Sham WMT + Sham rTMS
Number analyzed (Participants) | 11 | 9 | 10 | 11
units on a scale | -.113 (.426) | .091 (.133) | .208 (.256) | .197 (.376)

ADVERSE EVENTS:
Time Frame: The time frame was approximately 4 weeks, from the baseline study visit, throughout the treatment application period, until the final outcome assessment.
Description: Definitions do not differ from clinicaltrials.gov definitions.
Arm/Group | WMT + rTMS | Sham WMT + rTMS | WMT + Sham rTMS | Sham WMT + Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/12 | 1/9 | 0/11 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WMT + rTMS (N=12) | Sham WMT + rTMS (N=9) | WMT + Sham rTMS (N=11) | Sham WMT + Sham rTMS (N=11)
Discomfort during stimulation session. (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — Discomfort during stimulation session (head pain, tingling)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT03337113/Prot_SAP_ICF_000.pdf